CLINICAL TRIAL: NCT04039542
Title: A Mixed Methods Feasibility Study of a Transdiagnostic Compassion Focused Therapy (CFT) Group for Older Adults
Brief Title: A Feasibility Study of a Transdiagnostic Compassion Focused Therapy (CFT) Group for Older Adults
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 restrictions limited recruitment
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GN19MH088
Record Dates: First submitted 2019-07-01; First posted 2019-07-31 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: Depression; Anxiety Disorders
Keywords: Feasibility; Compassion Focussed Therapy; Older adults
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Mixed methods - qualitative and quantitative
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Compassion focused therapy (CFT) (Experimental): A group programme of CFT running for 10 sessions lasting 90 minutes per session.
  Interventions: Other: Compassion focused therapy (CFT)

INTERVENTIONS:
Other: Compassion focused therapy (CFT) — Compassion focused therapy (CFT) sessions (developed from cognitive behavioural therapies) to target underlying shame and self-criticism - 10 x 90 minute sessions

SUMMARY:
Compassion focused therapy (CFT) is a relatively new psychological therapy. Research has shown that CFT can improve psychological wellbeing and functioning in people with anxiety and depressive disorders. Research into CFT has focused on working age adults. It would be useful to evaluate whether CFT could be of benefit to the older adult population.

The present study aims to use the Medical Research Council (MRC) framework for developing and evaluating new treatments for complex conditions such as mental health. The present study aims to explore the feasibility and acceptability of a CFT group as a treatment for older adults with anxiety or depressive disorders. Additionally, the study aims to use the statistical data to inform future research.

Participants will be older adults (aged 60+) referred to National Health Service (NHS) Greater Glasgow and Clyde (GGC) older people's mental health service for common mental health conditions. People with psychosis, addictions, diagnosis of dementia or risk of self-harm will be ineligible. Participants will be offered the group as part of their treatment. Participants in the group will be identified and approached by an NHS clinician and asked to consent to participate in the study; non participation in the study will not affect their place in the group. The group protocol has been developed from previous research and will last for 10 weekly sessions of 90 minutes.

The study is mixed methods, using both quantitative and qualitative data. The quantitative part will use outcome measures which will look for a statistical relationship between the CFT group and changes in wellbeing and functioning. The qualitative part will use a semi-structured interview to hear people's experiences.

The CFT group will be delivered by an NHS clinical psychologist and Community Psychiatric Nurse (CPN).

DETAILED DESCRIPTION:
Recruitment Procedure:

Potential participants will be recruited from the older adult service within NHS GGC. Multidisciplinary team (MDT) staff within the service will identify potential participants for a CFT group and if they agree to participate in the group, attendees will then be asked to participate in the study by the student researcher. Group attendees' inclusion in the group is not dependent on their participation in the study. Inclusion and exclusion criteria will be assessed by Principal Clinical Psychologist and eligible participants will be asked for their consent to participate in the project by Trainee Clinical Psychologist.

Outcome Measures:

Principal Clinical Psychologist will administer outcome measures at beginning and end of the group programme. Additionally, measures will be administered after specific sessions to assess the effect of specific interventions.

Outcome measures to be used are -

Clinical Outcomes:

* Patient Health Questionnaire (PHQ-9) - a 9 item self-report measure of depressive symptoms.1 minute completion time. Administered after sessions 1, 5, 10.
* Generalized Anxiety Disorder (GAD-7) - a 7 item self-report measure of anxiety symptoms. 1 minute completion time Administered after sessions 1, 5, 10.

Mechanisms of Change:

• Forms of self-criticising/attacking & self-reassuring scale (FSCRS) - a self-report measure of self-criticism and self-reassurance. Used to evaluate the level of self-criticism a person experiences, which is often linked to mental health problems. Additionally, it evaluates the ability to reassure oneself. 4 minutes completion time.

Administered after sessions 1, 9, 10.

* Self-compassion scale (SCS) - a self-report measure measures a person's ability to show themselves compassion in the face of challenges. 4 minutes completion time. Administered after sessions 1, 8, 10.
* Toronto Mindfulness Scale - Trait - a self report measure of mindfulness traits such as curiosity, acceptance and openness. Given the CFT group incorporates elements of mindfulness, this will be useful to measure. 3 minutes completion time. Administered after sessions 1, 7, 10.
* Other as Shamer Scale - a self-repost measure to evaluate beliefs a person has about other's evaluation of them. 3 minutes completion time. Administered after sessions 1, 5, 10.
* Social Connectedness Scale - Revised - a self-report measure which evaluate people's feelings of connectedness to others. To measure whether the group itself has an impact on people's feelings. 4 minutes completion time. Administered after sessions 1, 5, 10.

Design:

As this is a feasibility study, a mix methods study design will be used. For the quantitative part of the study a within group design will be used to assess outcomes at baseline and posttreatment. Treatment acceptability will also be evaluated by semi-structured interviews following the intervention.

CFT Protocol:

A group programme of CFT will run for 10 sessions lasting 90 minutes per session. The group has been developed by an experienced NHS Clinical Psychologist working with older adults. The group protocol has been developed from a previous group run in NHS GGC with working age adults. The group will be delivered by NHS clinicians and led by Dr John Hickey. The sessions are titled as follows:

Session 1: Introduction, aims and soothing rhythm breathing Session 2 & 3: Psychoeducation Session 4: Formulation Session 5: Formulation & the threat system Session 6: Compassionate Self Session 7: Compassionate Image and barriers to compassion Session 8: Multiple selves - responding with different emotions Session 9: Shame and self-criticism Session 10: Review, formulation and planning ahead Participants will be asked to practice techniques and record their progress throughout the intervention. They will practice breathing and mindfulness techniques and keep a compassionate diary to support their learning.

Data Collection:

All outcome measures will be completed by participants pre-intervention, they will be posted to participants prior to the group (once consent has been received) and they will be asked to bring them to the first session. Copies will be available at the first session in case participants forget to bring them or have difficulties completing them. Time will be available to complete measures if necessary. The measures will also be repeated after specific sessions to evaluate any change from a specific intervention. Demographic data will also be obtained to allow for a description of the data.

The lead clinician will administer and collect the outcome measures at the end of the specified session. Attendance and dropout from the group will also be recorded for analysis.

Following the completion of the group, participants will be asked to attend for a semi-structured interview to discuss their experience of the CFT group protocol. All those who consented to participate in the study will be asked to participate in the semi-structured interview. The interviews will be conducted by Fiona McConnell (Trainee Clinical Psychologist). Interviews will be based on a topic guide, which will focus on the participant's experience of the intervention and their thoughts for improvements. The interviews will be audio recorded and transcribed and all patient identifiable data will be anonymised. The recordings will be destroyed once the project is complete.

ELIGIBILITY:
Inclusion Criteria:

* Experiencing symptoms of depression and/or anxiety disorder
* Able to provide informed consent
* English fluency

Exclusion Criteria:

* Psychosis
* Addictions
* Cognitive impairment
* Risk of self-harm

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-06-19 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Depressive symptoms | Baseline, 5 weeks and 10 weeks
  Change in Patient Health Questionnaire (PHQ-9) score: 9 item self-report measure. Scale range 0-27; higher score indicates increase in depression symptoms (worse)
Anxiety symptoms | Baseline, 5 weeks and 10 weeks
  Change in Generalized Anxiety Disorder (GAD-7) score: 7 item self-report measure. Scale range 0-21; higher score indicates increase in anxiety symptoms (worse)

SECONDARY OUTCOMES:
Self-criticism/self-reassurance | Baseline, 9 weeks and 10 weeks
  Change in Forms of self-criticising/attacking & self-reassuring scale (FSCRS) score: inadequate self sub-scale. Scale range 0-36; higher score indicates an increase in feelings of personal inadequacy (worse)
Self-criticism/self-reassurance | Baseline, 9 weeks and 10 weeks
  Change in Forms of self-criticising/attacking & self-reassuring scale (FSCRS) score: hated self sub-scale. Scale range 0-20; higher score indicates an increase in feelings of desire to persecute oneself (worse)
Self-criticism/self-reassurance | Baseline, 9 weeks and 10 weeks
  Change in Forms of self-criticising/attacking & self-reassuring scale (FSCRS) score: reassured self sub-scale. Scale range 0-32; higher score indicates an increase in feelings of ability to reassure oneself (better)
Self-compassion | Baseline, 8 weeks and 10 weeks
  Change in Self-compassion scale (SCS) total score. Scale range 0-130; higher score indicates an increase in feelings of self-compassion (better)
Mindfulness traits | Baseline, 7 weeks and 10 weeks
  Change in Toronto Mindfulness Scale - Trait score. Scale range 0-52; higher score indicates an increase in experiences of mindfulness (better)
Belief of others' evaluation | Baseline 5 weeks and 10 weeks
  Change in Other as Shamer Scale score. Scale range 0-72; higher score indicates an increase in feelings of external shame (worse)
Social connectedness | Baseline, 5 weeks and 10 weeks
  Change in Social Connectedness Scale - Revised score. Scale range 8-48; higher score indicates more social connectedness (better)

CONTACTS AND LOCATIONS:
Overall Officials: Hamish McLeod, PhD, Study Chair — University of Glasgow
Locations (1):
- NHS Greater Glasgow and Clyde, Glasgow, United Kingdom